CLINICAL TRIAL: NCT07370376
Title: Ultrasonographic Assessment of Diaphragmatic Function in Obstructive Sleep Apnea Patients
Brief Title: Ultrasonographic of Diaphragmatic Function in Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MohamedAbdElmoniem, Lecturer of chest medicine, Mansoura University
Other Study IDs: MS.23.03.2352
Record Dates: First submitted 2026-01-10; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: OSA
Keywords: Ultrasonographic Assessment; Diaphragmatic Function; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — 30 newly diagnosed OSA patients (AHI ≥5) and 30 age- and sex-matched non-OSA controls (AHI <5) were included. Exclusion criteria included systemic organ failure, uncontrolled diabetes, chronic respiratory diseases, neuromuscular disorders, prior OSA treatment, and steroid use. All participants underwent pulmonary function testing, and completed Epworth Sleepiness Scale (ESS), Berlin, and STOP-Bang questionnaires. Overnight, attended polysomnography (PSG) was performed following AASM guidelines. Diaphragm ultrasonography measured excursion, thickness at end-expiration and inspiration, and diaphragm thickening fraction (DTF).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- newly diagnosed OSA patients (AHI ≥5): 30 newly diagnosed OSA patients (AHI ≥5). All participants underwent pulmonary function testing, and completed Epworth Sleepiness Scale (ESS), Berlin, and STOP-Bang questionnaires. Overnight, attended polysomnography (PSG) was performed following AASM guidelines. Diaphragm ultrasonography measured excursion, thickness at end-expiration and inspiration, and diaphragm thickening fraction (DTF).
- non-OSA controls (AHI <5): All participants underwent pulmonary function testing, and completed Epworth Sleepiness Scale (ESS), Berlin, and STOP-Bang questionnaires. Overnight, attended polysomnography (PSG) was performed following AASM guidelines. Diaphragm ultrasonography measured excursion, thickness at end-expiration and inspiration, and diaphragm thickening fraction (DTF).

SUMMARY:
Obstructive sleep apnea (OSA) is associated with altered respiratory mechanics, including diaphragmatic function. Ultrasonography provides a non-invasive tool to assess diaphragmatic structure and performance, which may correlate with OSA severity.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is associated with altered respiratory mechanics, including diaphragmatic function. Ultrasonography provides a non-invasive tool to assess diaphragmatic structure and performance, which may correlate with OSA severity. The aim of the study is to evaluate diaphragmatic function in OSA patients using ultrasonography and to investigate its relationship with OSA severity and sleep-related parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting the Sleep Disordered Breathing (SDB) Unit at the Chest Medicine Department and diagnosed with obstructive sleep apnea (OSA) were included if they met the following criteria:
* Age 18-65 years.
* Willingness to participate in the study.

Exclusion Criteria:

* Patients were excluded if they had any of the following conditions:
* Refusal to participate in the study
* Age <18 or >65 years
* Systemic organ failure, including heart failure, stroke, renal failure, or liver failure; Uncontrolled diabetes mellitus
* Diagnosed obesity hypoventilation syndrome (OHS) or other sleep disorders apart from OSA
* Chronic respiratory diseases such as COPD, bronchial asthma, or restrictive lung disease
* OSA patients already receiving therapy (CPAP, oral appliances, or upper airway surgery)
* Neuromuscular disorders or other conditions affecting diaphragmatic function (malnutrition, chest trauma, or immobility)
* Use of steroids or uncontrolled autoimmune diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients visiting the Sleep Disordered Breathing (SDB) Unit at the Chest Medicine Department and diagnosed with obstructive sleep apnea (OSA) were included if they met the following criteria: Age 18-65 years.; OSA group: Newly diagnosed OSA confirmed by full-night polysomnography (PSG) with apnea-hypopnea index (AHI) > 5 events/hour; Control group: Patients with AHI < 5 events/hour on PSG; Willingness to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Assessment of Diaphragmatic Function in Obstructive Sleep Apnea Patients | 6 months
  All participants underwent diaphragm thickening fraction (DTF) as a percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Lecturer of chest medicine faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt